CLINICAL TRIAL: NCT01138839
Title: Dexamethasone Efficacy in HELLP I Syndrome, a Multicentric, Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Dexamethasone Efficacy in HELLP I Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Responsible Party: Javier Fonseca, Universidad del Valle
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1625; COLCIENCIAS RC No. 334-2008 (Other: colciencias)
Record Dates: First submitted 2010-05-10; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: HELLP Syndrome
Keywords: HELLP 1; Dexamethasone; Clinical trial
MeSH Terms: conditions — HELLP Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sterile water (Placebo Comparator): Pregnant women will receive 2.5 cc of sterile water every 12 hours until delivery and 3 additional doses after delivery. Puerperal women will receive 3 doses after delivery.
  Interventions: Drug: sterile water
- Dexamethasone (Experimental): Pregnant women in the experimental group will receive 10-mg doses (2.5 cc) of dexamethasone sodium phosphate intravenously every 12 hours until delivery and 3 additional doses after delivery. Puerperal women will receive 3 10-mg doses after delivery.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Pregnant women in the experimental group will receive 10-mg doses (2.5 cc) of dexamethasone sodium phosphate intravenously every 12 hours until delivery and 3 additional doses after delivery. Puerperal women will receive 3 10-mg doses after delivery.
  Other Names: steroid ev
  Arms: Dexamethasone
Drug: sterile water — Pregnant women will receive 2.5 cc of sterile water every 12 hours until delivery and 3 additional doses after delivery. Puerperal women will receive 3 doses after delivery
  Arms: sterile water

SUMMARY:
The purpose of this study is to determine the efficacy of dexamethasone for treatment of HELLP I (hemolysis, elevated liver enzymes and low platelet count) syndrome.

DETAILED DESCRIPTION:
Treatment of HELLP syndrome usually is restricted to measures of support and treatment of complications. In 2005, in a subgroup analysis we showed that, among patients with HELLP 1, there were a shorter average time to platelet recovery and less duration of hospitalization in women who received dexamethasone therapy, however the importance of this finding is diminished because this was an unplanned analysis and the severity of the disease was not taken into account at randomization.

ELIGIBILITY:
Inclusion Criteria:

* Women who were at >20 weeks of gestation or during the first 3 days of puerperium if hypertension developed during the pregnancy or the puerperium with:
* platelet count, < or = 50,000/mm3; aspartate aminotransferase (AST), > or = 70 U/L; lactate dehydrogenase (LDH), > or = 600 U/L.
* Women who consent to be included informed consent by signature

Exclusion Criteria:

* diabetic ketoacidosis
* oral temperature > 37.5 grade
* Contraindication for use steroids

Ages: 10 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization | Average: 15 days

SECONDARY OUTCOMES:
Recovery time of platelets to more than 100000/mm3 | Average:7 days
Recovery of AST, ALT and LDH | Average: 10 days
Transfusion of blood products | Average: 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Javier Fonseca, Dr, Principal Investigator — Universidad del Valle
Locations (1):
- Universidad del Valle, Cali, Valle del Cauca Department, Colombia